CLINICAL TRIAL: NCT05787730
Title: Ultrasound and Cure Rate Three Months and 15 Years After TOT-procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: T283/2022
Record Dates: First submitted 2023-02-20; First posted 2023-03-28 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Urinary Incontinence,Stress
Keywords: TOT; Perineal ultrasound
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients operated with TOT (Other): The study is a retrospective cohort study. Between 2005 and 2008, a total of 54 patients were examined with ultrasound before and after TOT surgery. The collected data has not been previously published. Now these same patients are to be examined again with a more advanced ultrasound device.
  Interventions: Device: Transobturator tape

INTERVENTIONS:
Device: Transobturator tape

SUMMARY:
The study is a cohort study. Between 2005 and 2008, a total of 54 patients were examined with ultrasound before and after TOT surgery. The collected data has not been previously published. Now these same patients are to be examined again with a more advanced ultrasound device.

The subjects underwent a urogynecological ultrasound examination before surgery and during the follow-up examination 2-3 months after the procedure. In connection with the follow-up examination, the success of the procedure and the satisfaction of the patients have been evaluated. The data was collected between 2005 and 2008, and the purpose is to invite the patients in question to a research visit, so that the long-term effect of the procedure can be evaluated and the position of the band can be determined with a newer technology ultrasound device. The patients' subjective satisfaction with the procedure is assessed using questionnaires.

DETAILED DESCRIPTION:
The study is a retrospective cohort study. Between 2005 and 2008, a total of 54 patients were examined with ultrasound before and after TOT surgery. The collected data has not been previously published. Now these same patients are to be examined again with a more advanced ultrasound device.

The study's inclusion criterion has been stress or mixed incontinence, for which surgical treatment has been indicated. The cough test must have been positive with a 300 ml bladder filling and the separation points <7 in the incontinence charts.. Exclusion criteria included previous incontinence surgery, simultaneous other gynecological surgery, residual urine volume >100 ml, lower urinary tract anomaly, urinary tract infection, more than three urinary tract infections per year, more than second-degree gynecological organ deposition, BMI >35, previous pelvic radiation therapy or active malignancy. Patients with anticoagulant therapy, anticholinergic or duloxetine medication, hemophilia or neurological disease that could cause bladder dysfunction were also not included in the study. Patients who did not understand the importance of research and treatment or who were unable to exercise were also not suitable for the study.

The subjects underwent a urogynecological ultrasound examination before surgery and during the follow-up examination 2-3 months after the procedure. In connection with the follow-up examination, the success of the procedure and the satisfaction of the patients have been evaluated. The data was collected between 2005 and 2008, and the purpose is to invite the patients in question to a research visit, so that the long-term effect of the procedure can be evaluated and the position of the band can be determined with a newer technology ultrasound device. The patients' subjective satisfaction with the procedure is assessed using questionnaires.

The research visit is carried out at Tyks' Gynecology Outpatient Clinic. During the research visit, the subject is subjected to a gynecological clinical examination, which includes a cough test, and a urogynecological ultrasound examination. Prior to the study visit, the subject is provided with written information about the study and questionnaire forms, which the patient brings with her to the study visit. Written consent to the study has been requested from all women participating in the study. Now the subjects will be asked for their consent again. Permission for the research has been requested from the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Has been stress or mixed incontinence, for which surgical treatment has been indicated.
* The cough test must have been positive with a 300 ml bladder filling
* The separation points <7 in the incontinence charts

Exclusion Criteria:

* previous incontinence surgery
* simultaneous other gynecological surgery
* residual urine volume >100 ml
* lower urinary tract anomaly
* urinary tract infection
* more than three urinary tract infections per year
* more than second-degree gynecological organ deposition
* BMI >35
* previous pelvic radiation therapy or active malignancy.
* Patients with anticoagulant therapy
* hemophilia or neurological disease that could cause bladder dysfunction

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Subjective cure | 15 years after operation
  Subjective cure is defined if patient answer to be very satisfied or satisfied with the TOT-procedure
Objective cure | 15 years after operation
  The cough stress test is negative performed in a semilithotomy position with a comfortably filled bladder (200-300 ml)

IPD SHARING:
Plan to Share IPD: No